CLINICAL TRIAL: NCT00214929
Title: Cooperative Investigation Plan for Home Treatment of Pulmonary Embolism
Brief Title: Home Treatment of Pulmonary Embolism
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Carlos III Health Institute (Other Government)
Collaborators: Spanish Society of Pneumology and Thoracic Surgery (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PIO30192
Record Dates: First submitted 2005-09-16; First posted 2005-09-22 (Estimated); Last update posted 2005-12-09 (Estimated); Status verified 2005-08

CONDITIONS: Pulmonary Embolism
Keywords: Pulmonary Embolism; Therapy; Home Nursing; Economics
MeSH Terms: conditions — Pulmonary Embolism

INTERVENTIONS:
Behavioral: treatment at home

SUMMARY:
The best management in selected patients of pulmonary Embolism (PE) should be at home. The efficacy and safety treatment´s at home versus at hospital should be similar and quality of life should be better. Our purpose is to demostrate that Low weight molecular heparin (LWMH) at home for PE is at least as effective and safe at home as at hospital

DETAILED DESCRIPTION:
In order to carry out the Cooperative Investigation Plan for home treatment of pulmonary embolism, a network of multidisciplinary groups was built with the participation of 10 groups, distributed in 6 different regions and integrated within the Spanish Society of Pneumology and Thoracic Surgery (SEPAR).

Those groups will share a database integrated in the Spanish Registry on Thromboembolic Disease (RIETE), which is a project already being carried out and in which many of the groups of the network already participate.

The research project will be a study developed in two phases. In the first phase, predictive profiles for a favourable progression of the disease in patients with pulmonary embolism will be studied using the actual management of the disease with the current assistance model.

In the second phase, a randomized study comparing the efficacy and safety of two models of home treatment ( discharge from hospital during the first 72 hours after the diagnosis of PE and discharge from hospital during the first 5 days) in patients previously selected, according to predefined criteria which were modified on the basis of the results of phase I versus the current assistance model will be developed

The results will be measured in terms of efficacy, safety, economic burden, and quality of life in both models (at home and at hospital).

ELIGIBILITY:
Inclusion Criteria:

* The consecutive outpatients subjects diagnosed of PE at 10 different Spanish hospitals.
* A score of 2 or under in our prediction rule (risk score for short-term)
* Signed written Informed consent

Exclusion Criteria:

* A score over 2 in our prediction rule
* Patients with a PE requiring thrombolysis or surgical thrombectomy
* Patients with right ventricular dyskinesia in echocardiography at 48 hours from heparin therapy. (It is not necessary echocardiography for the model of discharge at 5 days)
* Troponin level over 0,1 g/L
* Patiens requiring oxygen therapy or under 93% in oxygen saturation level.
* Patients requiring intravenous analgesic therapy
* Patients with some medical or surgical conditions requiring to stay at hospital
* Patients with advanced chronic cardiovascular diseases (dyspnea III-IV NYHA)
* Patients with advanced chronic respiratory diseases (several COPD criteria of GOLD with FEV1< 50%)
* Documented congenital or acquired bleeding tendency /disorder (s)
* Documented current ulceration or angiodysplastic gastrointestinal disease
* Hemorrhagic stroke or recent (< 3 months prior to randomization) brain, spinal, or ophthalmological surgery.
* Recent surgery < 3 days
* Pregnancy
* Several Obesity (CMI over 30)
* Patients could not complete the treatment at home.
* Exclusion criteria related to study procedures
* Life expectancy < 3 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2004-12; Study Completion 2005-08

PRIMARY OUTCOMES:
-Thromboembolic recurrences
-Bleeding Complications
-Deaths

SECONDARY OUTCOMES:
-Quality of life

CONTACTS AND LOCATIONS:
Overall Officials: Remedios Otero, MD, Study Chair — Pneumology Service of Virgen de Rocio Hospital (Spain); Fernando Uresandi, MD, Principal Investigator — Pneumology Service.Cruces Hospital (Spain); David Jimenez, MD, Principal Investigator — Pneumology Service. Ramon y Cajal Hospital (Spain); Miguel A. Cabezudo, MD, Principal Investigator — Pneumology Service. H. Asturias (Spain); Francisco Conget, MD, Principal Investigator — Pneumology Service. Clinic Hospital of Zaragoza (Spain); Dolores Nauffal, MD, Principal Investigator — Pneumology Service. La Fe Hospital (Spain); Mikel Oribe, MD, Principal Investigator — Pneumology Service. Galdakao Hospital (Spain); Jose L. Lobo, MD, Principal Investigator — Pneumology Service. Txagorritxu Hospital (Spain); Fulgencio Gonzalez, MD, Principal Investigator — Pneumology Service. 12 de Octubre Hospital (Spain); Elena Laserna, MD, Principal Investigator — Pneumology Service. S.Juan de Dios Hospital (Spain)
Locations (1):
- Pneumology Service of HVR, Seville, Seville, Spain

REFERENCES:
- [Derived] Otero R, Uresandi F, Jimenez D, Cabezudo MA, Oribe M, Nauffal D, Conget F, Rodriguez C, Cayuela A. Home treatment in pulmonary embolism. Thromb Res. 2010 Jul;126(1):e1-5. doi: 10.1016/j.thromres.2009.09.026. Epub 2009 Oct 24. PMID 19853892
- See also: The clinical variables have been collected from the Spanish Computerized Registry of Patients with Venous Thromboembolism (R.I.E.T.E.) (www.riete.org) — http://www.riete.org